CLINICAL TRIAL: NCT02371564
Title: High Flow Oxygen Therapy in Patients Suffering From Chronic Obstructive Pulmonary Disease Exacerbation: Effects and Mechanisms of Action
Acronym: Oh BPCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHU-P 2013-25
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: COPD Exacerbation

ARMS (2):
- High flow humidified oxygen first (Active Comparator): High flow humidified oxygen then standard oxygenotherapy with a two-hour non invasive ventilation session in between.
  Interventions: Device: High flow humidified oxygen
- Standard oxygen therapy first (Active Comparator): Standard oxygenotherapy then high flow humidified oxygen with a two-hour non invasive ventilation session in between.
  Interventions: Device: Standard flow humidified oxygen

INTERVENTIONS:
Device: High flow humidified oxygen
  Arms: High flow humidified oxygen first
Device: Standard flow humidified oxygen
  Arms: Standard oxygen therapy first

SUMMARY:
Acute exacerbation of chronic obstructive pulmonary disease (COPD) is associated with poor outcome, especially when intubation is required, thus underlining the importance of optimizing non-invasive ventilatory support to avoid intubation. Practically, because of treatment intolerance, non-invasive ventilation (NIV) cannot be administered 24-hour a day for a long period of time and alternative solutions must be found to deliver oxygen as efficiently as possible to allow NIV interruptions. High flow humidified oxygen therapy (HFHO) consists of delivering a high-flow (15-60 L/minute) heated air-oxygen mixture (FIO2 21-100%) through a dedicated nasal cannula and can be interesting in this context. This well tolerated technique improves oxygenation and decreases respiratory rate and dyspnea in patients suffering from acute hypoxemic respiratory failure. In chronic COPD patients, using HFHO can decrease respiratory rate and PaCO2. In COPD exacerbation, using HFHO can conceptually be interesting. First, the high air-oxygen flow delivered well matches the patient's inspiratory demand and should decrease the work of breathing. Second, as during HFHO a high flow is continuously delivered in the airways, a wash-out of the anatomical dead space should occur and CO2 clearance should be enhanced. Despite this strong physiological rational for the use of HFHO in patients suffering from COPD exacerbation, the effects of using HFHO instead of conventional oxygenotherapy in combination with non-invasive ventilation (NIV) in this context has never been explored.

The main objective of the study is to explore the effects of using HFHO in combination with NIV in acute COPD exacerbation and to assess the underlying mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients suffering from acute hypercapnic respiratory failure (PaCO2 > 50 mmHg) due to COPD exacerbation and requiring intermittent NIV treatment can be included in the study provided they do not require immediate intubation.

Exclusion Criteria:

* Patients younger than 18 years old
* Inability to give informed consent or denied informed consent
* Severe acute respiratory failure requiring immediate intubation defined as respiratory rate > 40/minute, severe hypoxemia with PaO2/FIO2 ratio < 150 mmHg despite high FIO2, severe respiratory acidosis with pH< 7.2, altered mental status)
* Very intensive NIV treatment required defined as an impossibility to stop NIV treatment during more than one hour.
* Severe hypoxemia requiring more than 4l/minute of conventional oxygenotherapy between NIV treatments
* Poor short term prognosis (defined by the clinician in charge as a high risk of death during the next 7 days) or ongoing palliative treatment.
* Patients with "Do not resuscitate" order already established

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
corrected minute ventilation | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Angers, Angers, France